CLINICAL TRIAL: NCT00629668
Title: Genetic Polymorphisms of TNF-α Promoter and HBV Genotype on Outcome of HBV-Related Chronic Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KMUH-IRB-940189
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2007-07

CONDITIONS: Chronic Liver Disease; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Tumor Necrosis Factor-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: TNF-alpha and HBV genotype
Other: TNF-alpha and HBV genotypes

SUMMARY:
The prognosis of Hepatitis B virus (HBV)infection varies from minimal progressive liver disease to cirrhosis or hepatocellular carcinoma (HCC).Both viral and host genetic factors contribute to disease severity. Cytokine gene polymorphism has been regarded affecting prognosis of disease. By detecting HBV genotyping and tumor necrosis factor-alpha polymorphism, this study aime to assess their effects and interaction on disease severity of HBV-related chronic liver disease and HCC.

ELIGIBILITY:
Inclusion Criteria:

* HBV-positive patients

Exclusion Criteria:

* HBV-negative patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-01; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
cytokine gene polymorphism | years

SECONDARY OUTCOMES:
cytokine gene polymorohism on severity of disease | years

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Eing Jeng, M.D., Principal Investigator — Assistant Professor of Clinical Laboratory
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan